CLINICAL TRIAL: NCT03154385
Title: RITUX-PLUS. A Prospective Open Trial to Assess the Efficacy and Safety of a Treatment Combining Rituximab and Belimumab in Adults With Persistent Immune Thrombocytopenia.
Brief Title: Efficacy and Safety Assessment of a Treatment Combining Rituximab and Belimumab in Adults With Persistent Immune Thrombocytopenia
Acronym: RITUX PLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P130408
Record Dates: First submitted 2017-04-13; First posted 2017-05-16 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab; belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- arm 1 (Experimental): Two intravenous perfusions of 1 g of Rituximab (Mabthera ®) at W0 and W2 coupled with 100 mg intravenous methylprednisone to avoid potential allergic reactions.
  Five belimumab (Benlysta ®) injections will be administered (W0 + 2days, W2 + 2 days, W4, W8, W12) at 10mg/kg doses. The first two injections are administered 2 days after Rituximab perfusions. The adopted experimental scheme was once used to show use of belimumab in systemic lupus erythematosus in accordance with AMM regulation
  Interventions: Drug: Rituximab (Mabthera ®) Belimumab (Benlysta ®)

INTERVENTIONS:
Drug: Rituximab (Mabthera ®) Belimumab (Benlysta ®) — Rituximab (Mabthera ®): 1g IV at W0 and W2 Belimumab (Benlysta ®) : 10mg/kg IV, W0 + 2days, W2 + 2 days, W4, W8, W12

SUMMARY:
Previous studies have shown that increase level of BAFF could promote the settlement of long-lived plasma cells in the spleen of ITP patients treated with anti-CD20. This single-center prospective pilot study, currently in phase IIa, will evaluate the efficacy of a rituximab and belimumab sequential combination treatment. Investigators plan to include 15 patients with persistent ITP over a 24-month inclusion period. Each patient will be followed for 1 year

DETAILED DESCRIPTION:
This single-center prospective pilot study, currently in phase IIa, evaluates the efficacy of a rituximab and belimumab sequential combination treatment. Based on the Fleming method, this study scheme includes a single step method.

Eligible patients, having given consent and having been verified for inclusion criteria, will receive two intravenous perfusions of 1 g of Rituximab (Mabthera ®) at W0 and W2 coupled with 100 mg intravenous methylprednisone to avoid potential allergic reactions.

Five belimumab (Benlysta ®) injections will be administered (W0 + 2days, W2 + 2 days, W4, W8, W12) at 10mg/kg doses. The first two injections are administered 2 days after Rituximab perfusions. The adopted experimental scheme was once used to show use of belimumab in systemic lupus erythematosus in accordance with AMM regulation.

This phase II prospective single-center open-trial will be conducted at the National Referral Center for Adult Immune Cytopenia located in the Henri Mondor University Hospital. Investigators plan to include 15 patients with persistent ITP over an 24-month inclusion period. Each patient will be followed for 1 year

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, <75 years
* Primary ITP diagnostic defined according to the standard definition criteria (Rodeghiero et al Blood 2008)
* Previous transient response to first-line treatments of corticosteroids and/or IgIV characterized by a rise of platelet levels > 30 G/L with at least a twofold increase from baseline levels followed by a relapse.
* Platelet count ≤ 30,000 /µL at inclusion or <50 G/L if presence of hemorrhagic events or other reason left up to investigator discretion.
* A persistent ITP active and existing for more than 3 months but less than 5 years from diagnosis.
* Normal Bone marrow smear for patients above 60 years of age
* Negative pregnancy test results for women of procreation age
* Gammaglobulin level > 7 g/L
* Informed consent

Exclusion Criteria:

* Splenectomy
* Previous treatment by Rituximab or any B-cell targeted therapy
* Previous treatment by cyclophosphamide
* No medical treatments of a therapeutic protocol nature within the last 30 days
* Previous anaphylactic shock
* Previous septic shock or severe sepsis
* Chronic and ongoing severe infection requiring treatment or hospitalization in the 60 days preceding inclusion.
* Severe acute infection within the last 4 weeks
* Use of parenteral antibiotics within 60 days current use of suppressive therapy for chronic infection such as tuberculosis, pneumocystis, cytomegalovirus, HSZ, herpes zoster, and atypical mycobacteria
* History of primary immunodeficiency, IgG level < 400 mg/dl and/or IgA level < 10 mg/dl
* Have evidence of serious suicide risk including any history of suicidal behavior in the last 6 months and/or any suicidal ideation in the last 2 months or who in the investigator's judgment, pose a significant suicide risk.
* Secondary ITP
* History of recurrent infections
* Neutrophils count < 1,000/mm3 at inclusion
* Positive HIV test and/or hepatitis virus C infection and/or positive hepatitis B virus surface antigen or core antibody (HbsAg or HBcAb)
* Impaired renal function as indicated by a serum creatinine level > 2 mg/dl
* New York Heart Classification III or IV heart disease
* Treatment by antiaggregant/antiplatelet or anti-vitamin K drug
* Previous history of malignancy in the last 5 years other than cutaneous carcinoma
* Previous history of severe psychiatric disorder or previous suicide attempts in the last 6 months or suicidal thoughts in the last 2 months leading up to inclusion
* Unable to comply with study and follow-up procedures due to psychiatric disorders or any other reason
* Alcohol or drug abuse or dependence, either current or within 1year
* Pregnancy or Breast-Feeding
* Live, attenuated vaccinations must be administered at least 30 days before inclusion in study
* History of significant medical illness or clinically significant laboratory abnormality (or planned surgical procedure) which in the opinion of the investigator would interfere with the study procedures and / or assessments or compromise subject safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
The total number of patient responses to treatment, in other words sum of complete responses + responders | Week 52
  A responder (R) to treatment is defined by a patient with a maintained platelet count at >30x109/L (Rodeghiero et al Blood 2008) and a minimum twofold increase from initial platelet levels in the absence of bleeding and/or use of ITP directed therapies between Week 6 and Week 52 of patient follow-up.
  A complete response (CR) is defined by a platelet count > 100 x 109/L maintained in the absence of any other ITP directed therapies between Week 6 and Week 52.
  A Non-Responder (NR) is a patient with one or all of the following :
  1. Platelet count less than < 30 x 109/L by the end of study
  2. Require a rescue therapy (a new course of corticosteroids and/or intravenous immunoglobulin) more than 6 weeks after inclusion.
  3. Underwent any other treatment for ITP over the study period

SECONDARY OUTCOMES:
Number of patients developing a severe hypogammaglobulinemia (gammaglobulin level < 4 g/dl) | at weeks 12, 24, 36, and 52
Evolution of gammaglobulin levels | at weeks 4, 8, 12, 24, 36, and 52
Duration of severe hypogammaglobulinemia in patients with such complication | Week 24
Variation in gammaglobulin subclass levels throughout the study | at weeks 0,12, 24, 36, 52
Number of severe infections requiring hospitalization | at weeks 24, 36 and 52
Platelet Levels | at weeks 4, 8, 12, 24, 36, and 52
Total number of responders (responders + complete responses) | at weeks 12,25, and 36

CONTACTS AND LOCATIONS:
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Derived] Mahevas M, Azzaoui I, Crickx E, Canoui-Poitrine F, Gobert D, Languille L, Limal N, Guillaud C, Croisille L, Jeljeli M, Batteux F, Baloul S, Fain O, Pirenne F, Weill JC, Reynaud CA, Godeau B, Michel M. Efficacy, safety and immunological profile of combining rituximab with belimumab for adults with persistent or chronic immune thrombocytopenia: results from a prospective phase 2b trial. Haematologica. 2021 Sep 1;106(9):2449-2457. doi: 10.3324/haematol.2020.259481. PMID 32817288